CLINICAL TRIAL: NCT02688348
Title: Prospective Study of Bladder-Preservation Chemo-Radiotherapy (Partial Bladder Hypo-fractionated Radiotherapy) for Patients With Muscle-Invasive Bladder Cancer
Brief Title: Quality of Life After Bladder-Preservation Chemotherapy and Radiation Therapy in Patients With Muscle-Invasive Bladder Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 15-000496; NCI-2015-01765 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); JCCCID556 (Other: Jonsson Comprehensive Cancer Center); 15-000496 (Other: UCLA / Jonsson Comprehensive Cancer Center)
Record Dates: First submitted 2016-02-10; First posted 2016-02-23 (Estimated); Last update posted 2020-07-24 (Actual); Status verified 2020-02

CONDITIONS: Infiltrating Bladder Urothelial Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ancillary-Correlative (late toxicity and QOL) (Other): Patients complete the EORTC QLQ-BLM-C30 at baseline, every 3 months for 1 year, every 4 months for 1 year, every 6 months for 3 years, and then annually thereafter after completion of chemo-radiotherapy.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This research trial studies quality of life after bladder-preservation chemotherapy and radiation therapy (chemo-radiotherapy) in patients with bladder cancer that has spread into or through the muscle layer of the bladder (muscle-invasive bladder cancer). Bladder-preservation chemo-radiotherapy is a standard treatment for patients with muscle-invasive bladder cancer, however, chemo-radiotherapy may cause urinary tract, bowel, and sexual late side effects that negatively affect patients' quality of life. Studying quality-of-life in patients with muscle-invasive bladder cancer after chemo-radiotherapy may help identify the long-term side effects of treatment and may help plan the best treatment in the future and improve patients' quality of life.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To study health-related quality of life (HRQoL, or QOL) for patients undergoing protocol-based bladder-preservation chemo-radiation.

OUTLINE:

Patients complete the European Organization for Research and Treatment for Cancer (EORTC) QLQ-Bladder Cancer Muscle Invasive (BLM-C30) at baseline, every 3 months for 1 year, every 4 months for 1 year, every 6 months for 3 years, and then annually thereafter after completion of chemo-radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed muscle-invasive urothelial cancer (no histology will be excluded)
* No pelvic nodal metastases or distant metastases (based on computed tomography [CT], positron emission tomography [PET] or magnetic resonance imaging [MRI])
* Karnofsky performance status (KPS) >= 70
* Ability to understand, and willingness to sign, the written informed consent
* Patient will have either opted for bladder-sparing treatment as compared to radical cystectomy, or deemed medically inoperable
* Following the recent recommendations from the International Consultation on Urological Diseases-European Association of Urology International Consultation on Bladder Cancer, eligible patients will be those with no hydronephrosis, no extensive carcinoma in situ (CIS), and no tumor invasion into the stroma of the prostate

Exclusion Criteria:

* Patients with any evidence of distant metastases
* Prior pelvic radiotherapy
* History of Crohn's disease or ulcerative colitis
* Unable to receive chemotherapy
* Histologies other than urothelial (eg. squamous cell carcinoma, adenocarcinoma, small cell)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-04-22 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Establish QOL with validated tools for patients undergoing bladder-preservation chemo-radiation | From the date of study entry up to 5 years
  Validated Quality-of-Life questionnaires developed by the European Organization for Research and Treatment for Cancer (EORTC) will be used. The EORTC QLQ-BLM30 with 30 questions specific to muscle-invasive bladder cancer will be combined and used in conjunction with the general cancer questionnaire EORTC QLQ-C30 (Aaronson).

SECONDARY OUTCOMES:
Quantify the rate of early and late grade 3 or higher GU or GI toxicity based on the CTCAE criteria | Up to 5 years
Overall survival | From the date of study entry to the date of death, assessed up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Christopher King, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States